CLINICAL TRIAL: NCT05318924
Title: Will Work for Reward: Effects of Ghrelin Administration on Dopamine and Effort
Brief Title: Effects of Ghrelin Administration on Dopamine and Effort
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: DFG KR 4555/7-1
Record Dates: First submitted 2022-02-22; First posted 2022-04-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder
Keywords: energy homeostasis; PET/MR; dopamine; motivation; ghrelin
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ghrelin

STUDY DESIGN:
Intervention Model Description: The investigators will assess the effects of intravenous administration of ghrelin on dopamine signaling using a double-blind randomized cross-over design. To this end, 26 healthy participants will be infused with ghrelin (vs. saline) while we determine dopamine release (via PET imaging) and assess cerebral blood flow and functional connectivity at rest (via concurrent MR imaging).
  These 26 healthy participants will be drawn from a larger sample of 100 participants (including 50 patients with major depressive disorders), who will complete a reward task battery that will be associated with fasting blood levels of ghrelin.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Neither participants nor investigators will know whether the participant receives a ghrelin or saline infusion, which will be prepared by independent members of the university hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ghrelin infusion (Experimental): To achieve approximately stable elevated ghrelin levels during the infusion procedure, the investigators will use a loading dose of 1 mcg/kg as well as an infusion rate of 0.051 mcg/kg/min in line with recent studies (Farokhnia, Grodin, Lee et al., 2017) and general recommendations (Garin, Burns, Kaul et al., 2013).
  Interventions: Drug: Ghrelin
- Placebo infusion (Placebo Comparator): Saline
  Interventions: Other: Placebo
- Patients with MDD (No Intervention): Patients with major depressive disorder will be enrolled for comparison to healthy participants on the reward task battery, but not randomized to the ghrelin vs. saline infusion.

INTERVENTIONS:
Drug: Ghrelin — Participants will receive an infusion that is intended to raise ghrelin level up to a steady plateau.
  Arms: Ghrelin infusion
Other: Placebo — Participants will receive a saline infusion as the placebo control condition.
  Arms: Placebo infusion

SUMMARY:
Ghrelin is a stomach-derived hormone and the only known circulating peptide that stimulates appetite. Animal studies have conclusively shown that ghrelin increases dopaminergic neurotransmission and, thereby, enhances effort. However, similar evidence on the putative role of ghrelin in humans is still lacking. Here, the investigators propose to conduct a [11C]-raclopride PET/MR study after intravenous administration of ghrelin vs. saline in healthy individuals. First, during an intake visit, the investigators will assess fasting blood levels of hormones involved in appetitive behavior such as ghrelin, leptin, and insulin. In addition, the investigators will conduct a set of tasks that have been associated with dopamine function (i.e., effort and reinforcement learning). Second, the investigators will assess the effects of intravenous administration of ghrelin on dopamine signaling using a double-blind randomized cross-over design. To this end, participants will be infused with ghrelin (vs. saline) while we determine dopamine release (via PET imaging) and assess cerebral blood flow and functional connectivity at rest (via concurrent MR imaging). Furthermore, the investigators will conduct an instrumental motivation task (IMT) where participants have to exert physical effort to obtain rewards. Based on preclinical studies and indirect evidence from human studies, the investigators hypothesize that ghrelin will increase dopamine release in the striatum and that this will, in turn, lead to an increase in the willingness to work for rewards. Moreover, the investigators expect that ghrelin-induced dopamine release will be associated with an elevated tracking of reward utility in the mesolimbic circuit during the IMT, which is known to be associated with response vigor. Collectively, the proposed project would provide a unique resource to test an important link between the gut and the brain in the regulation of appetitive behavior. If ghrelin were to enhance effort expenditure for rewards via dopamine signaling in humans, then restoring sensitivity to ghrelin might be the more promising therapeutic approach compared to antagonizing the ghrelin receptor.

ELIGIBILITY:
Inclusion Criteria:

* Healthy control participants: never fulfilled the criteria of any mood or anxiety disorder (except specific phobia)
* Patients with major depressive disorder: diagnosis according to DSM-5 within 12 months before enrollment and presence of at least mild symptoms at enrollment (BDI II >= 14)

Exclusion Criteria:

* lifetime history of a brain injury, schizophrenia, bipolar disorder, and a severe substance use disorder according to DSM-5
* obsessive-compulsive disorder, trauma- and stressor-related disorder, somatic symptom disorder, and eating disorder within a 12-month interval before the test day.
* Neuroimaging Study involving ghrelin infusion: contraindication for PET/MR (e.g., metal implants or prostheses, pregnancy, claustrophobia)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Ghrelin-induced changes in dopamine release | During the infusion (up to 90 min)
  [11C]raclopride binding potential after ghrelin infusion vs. saline infusion
Ghrelin-induced changes in motivation | During the infusion (60-90 min after start of the infusion)
  Force exerted on grip force controller to obtain rewards after ghrelin infusion vs. saline infusion
Ghrelin-induced changes in functional connectivity and perfusion | During the infusion (up to 90 min)
  Functional connectivity and perfusion of regions of the reward circuit (i.e., Nucleus Accumbens and Ventral Tegmental Area/Substantia Nigra) after ghrelin infusion vs. saline infusion
Changes (Ghrelin-induced) in hunger and satiety from baseline | Pre infusion and 20 minutes post infusion (compared to saline)
  Change in visual analogue scale (0-100) measures of subjective hunger and satiety after ghrelin infusion vs. saline infusion

SECONDARY OUTCOMES:
Ghrelin-induced changes in mood | Pre infusion and 20 minutes post infusion (compared to saline)
  Changes operationalized via visual analogue ratings (0-100) of positive and negative affect schedule mood items after ghrelin infusion vs. saline infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry & Psychotherapy, University of Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
After the publication of the key results of the study, all anonymized imaging data will be made publicly available (e.g., at openfmri.org). Behavioral data will be shared after aggregation at the trial or participant level.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available after an embargo period of 12 months after completion of the study.
Access Criteria: Until the data is publicly available, researchers may contact the lead PI to gain access.
URL: http://neuromadlab.org